CLINICAL TRIAL: NCT02667327
Title: A Phase 3, Randomized, Double-blind, Parallel-group, Vehicle Controlled, Multicenter Study of the Efficacy and Safety of Granexin Gel in the Treatment of Diabetic Foot Ulcer (GAIT 1)
Brief Title: A Study of Granexin Gel in the Treatment of Diabetic Foot Ulcer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision (No safety or efficacy concerns)
Sponsor: Xequel Bio, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-DFU-301; NCT02666131 (obsolete NCT alias)
Record Dates: First submitted 2016-01-26; First posted 2016-01-28 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Diabetic Foot Ulcers
Keywords: diabetic foot ulcer; diabetic complications; diabetes; wound healing; Granexin gel; FirstString Research
MeSH Terms: conditions — Diabetic Foot; Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Granexin gel plus Standard of Care (Active Comparator): Granexin gel is comprised of 100 μM aCT1 peptide plus hydroxyethyl cellulose.
  Interventions: Drug: Granexin gel
- Vehicle gel plus Standard of Care (Placebo Comparator): Vehicle gel is hydroxyethyl cellulose without active pharmaceutical ingredient.
  Interventions: Other: Vehicle gel
- Standard of Care (No Intervention): Standard of Care includes cleaning and irrigating ulcer, non-surgical debridement, pain management, ulcer dressing, off-loading, and nutritional assessment.

INTERVENTIONS:
Drug: Granexin gel — Granexin gel contains active pharmaceutical ingredient, aCT1 peptide, for topical application to diabetic foot ulcers once a week for up to 12 weeks or until wound closure, whichever comes first.
  Other Names: Granexin
  Arms: Granexin gel plus Standard of Care
Other: Vehicle gel — The vehicle gel formulation is hydroxyethyl cellulose that does not contain the active aCT1 peptide. Vehicle gel will be applied topically to diabetic foot ulcers once a week for up to 12 weeks or until wound closure, whichever comes first.
  Other Names: Control
  Arms: Vehicle gel plus Standard of Care

SUMMARY:
The purpose of this study is to determine whether Granexin gel is safe and effective in the treatment of diabetic foot ulcers.

DETAILED DESCRIPTION:
DFU patients will undergo a one week screening period and those with changes in ulcer size of less than 30% will be eligible for randomization providing all other criteria are met. Participants enrolled in the study will receive treatment based on randomization into 1 of 3 treatment arms for up to 12 weeks. The participants will have an additional 12 week follow-up period beyond the treatment period to assess durability of wound closure.

ELIGIBILITY:
Inclusion Criteria:

Both male and female participants may participate in the study.

To be eligible for entry into this study, a patient must meet all of the following Inclusion criteria:

1. Age 18 years or older
2. Established diagnosis of diabetes mellitus (type I or II)
3. Glycosylated hemoglobin (HbA1c) value < 12.0% at the screening visit
4. Diagnosis of neuropathic foot ulcer by 10g monofilament test, tuning fork (128 Hz), or cotton wisp
5. Designated foot ulcer meets the following criteria at both the screening and baseline visits:

   1. Present for at least 4 weeks
   2. Full-thickness cutaneous ulcer below the ankle surface
   3. University of Texas grade A1
   4. Wound area (after debridement) 1 to 40.0 cm2
   5. Viable, granulating wound (investigator discretion)
6. Ankle brachial index ≤ 0.7 at both the screening and baseline visits. If the ABI is >1.30, one of the following confirmatory tests must be performed for the patient to be considered eligible:

   1. Does Not have a monophonic or biphasic flow (with the loss of reverse flow) in the artery of the foot with the target ulcer via doppler waveform analysis of the dorsalis pedis and posterior tibial arteries, as determined by standard practices of the investigator and the site.
   2. Transcutaneous oxygen pressure (TcPO2) at the foot >40 mmHg

   Additionally, patients must meet all other protocol-defined eligibility criteria.
7. Signed informed consent
8. Female patients of childbearing potential must have a negative pregnancy test at screening and must agree to use hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence throughout until 2 weeks after the last administration of investigational product. Male patients must also agree to use contraception such as a condom.

Exclusion Criteria:

Patients will not be eligible for enrollment in the study if they meet any of the exclusion criterial listed below:

1. Change (decrease or increase) in size of the designated target ulcer by ≥ 30% during the 7-day screening period
2. Cannot tolerate the off-loading methods or cannot comply with study related procedures
3. Has an ulcer that meets any of the following criteria:

   1. Shows signs of severe clinical infection, defined as pus oozing from the ulcer site
   2. Requires surgical debridement
   3. Is positive for β-hemolytic streptococci upon culture performed prior to screening debridement procedure
   4. Has > 50% slough, significant necrotic tissue, bone, tendon, or capsule exposure
   5. Is highly exuding (i.e., requires daily change of dressing)
4. Requires total contact cast
5. Ankle brachial pressure index < 0.7
6. Has a local or systemic infection or local lymphangitis ≥ 0.5 cm
7. Has any 1 of the following (only 1 of the 2 tests is required):

   1. A monophasic or biphasic flow (with loss of reverse flow) in the artery of the foot with the target ulcer via doppler waveform analysis of the dorsalis pedis and posterior tibial arteries
   2. Transcutaneous oxygen pressure (TcPO2) at the foot <40 mgHg
8. Presence of active malignant or benign tumor of any kind, (with the exception to nonmelanoma skin cancer as per investigator's discretion)
9. Congestive heart failure (New York Heart Association class II-IV)
10. Coronary heart disease with ST segment elevation myocardial infarction or coronary artery bypass graft or percutaneous transluminal coronary angioplasty within the last 6 months
11. Active osteomyelitis of the foot with the target ulcer detected by x-ray, CT scan, or MRI
12. Active connective tissue disease
13. Acute or chronic Charcot's neuro-arthropathy as determined by clinical and/or radiographic examination
14. Active treatment with systemic corticosteroids or topical corticosteroids (for treatment of the target ulcer or any area of the foot). This does not include inhaled corticosteroids used for conditions other than treating the target ulcer or any area of the foot. Wash out period for systemic corticosteroids is 14 days for inclusion in this study. Wash out period for topical corticosteroids (for treatment of the target ulcer or any area of the foot) is 14 days for inclusion in the study)
15. Active treatment with systemic antibiotics (wash out period for systemic antibiotics is 7 days for the inclusion in the study)
16. Previous or current radiation therapy to the distal lower extremity or likelihood to receive this therapy during study participation
17. Pregnant or nursing mothers
18. Uncontrolled anemia (hemoglobin < 10 g/dL in females and < 12 g/dL in males)
19. Estimated glomerular filtration rate < 25 mL/min
20. Poor nutritional status, defined as an albumin < 25 g/L (< 2,500 mg/dl)
21. Significant peripheral edema as per investigator's discretion
22. Known inability or unavailability of a patient to complete required study visits during study participation
23. A psychiatric condition (e.g., suicidal ideation) or chronic alcohol or drug abuse problem, determined from the patient's medical history, which, in the opinion of the investigator, may pose a threat to patient compliance
24. Use of a platelet-derived growth factor within 28 days before screening
25. Use of any investigational drug or therapy within 28 days before screening
26. Has any other factor which may, in the opinion of the investigator, compromise participation and/or follow-up in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Incidence of complete wound closure at Week 12 based on investigator assessment | Week 12

SECONDARY OUTCOMES:
Time in days to first complete wound closure of the target ulcer based on investigator assessment over the 12 week treatment period | Week 12

CONTACTS AND LOCATIONS:
Locations (29):
- United States (6):
  - New Hope Podiatry Group, Inc., Los Angeles, California
  - Integral - Clinical Trials Solutions, Doral, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Nirvana Research Center, Miami, Florida
  - Acclaim Bone & Joint, Fort Worth, Texas
  - Futuro Clinical Trials, LLC, McAllen, Texas
- Centre podiatrique et soins des plaies, Boucherville, Quebec, Canada
- Hungary (2):
  - Clinexpert Kft. - Kaszasdulo utca 5., Budapest
  - Strazsahegy Medicina Bt., Zrinyi utca 226, Budapest
- India (16):
  - Shrey Hospital Pvt Ltd, Ahmedabad, Gujarat
  - Parul Sevashram Hospitals, Ahmedabad, Gujarat
  - Anand Multispecialty Hospital, Vadodara, Gujarat
  - Convenient Hospitals Ltd., CHL - Hospitals, Indore, Madhya Pradesh
  - KLEs Dr. Prabakar Kore Hospital and Medical Research Center, Belagavi
  - Peoples College of Medical Science and Research Centre, Bhopal
  - Marwari Hospital and Research Centre, Guwahati
  - Surakshaka MultiSpecialty and Diabetes Hospital, Hyderabad
  - KRM Hospital and Research Center, Lucknow
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow
  - Fortis Hospital, Mohali
  - K R Hospital and Research Institute, Mysore
  - Supe Heart and Diabetes Hospital and Research Centre, Nashik
  - Batra Hospital and Medical Research Center, New Delhi
  - Aman Hospital and Research Centre, Vadodara
  - Anu Hospitals, Kovelamudivara Street, Vijayawada
- Poland (4):
  - Instytut Medycyny Wsi - oddz diabetologii ul. Jaczewskiego 2, 20-090 Lublin, Poland, Lublin, Jaczewskiego
  - NZOZ MED ART. Poradnie Specjalistyczne Ks. Wladyslawa 27, 44-240 Zory, Poland, Żory, Wladyslawa 27
  - Lubuskie Centrum Diabetologii UI., Budziszynek, Zielon
  - MIKOMED Sp. z o.o. ul., Lodz, Łódź .Pługowa

IPD SHARING:
Plan to Share IPD: No